CLINICAL TRIAL: NCT00907062
Title: Ginkgo Biloba for the Treatment of Vitiligo Vulgaris in Adolescents: an Open Label Pilot Clinical Trial
Brief Title: Ginkgo Biloba for the Treatment of Vitiligo Vulgaris in Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Interdisciplinary Network Complementary & Alternative Medicine Research (Other)
Responsible Party: Heather Boon, Associate Professor, Leslie Dan Faculty of Pharmacy, University of Toronto
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHPD#-137767; REB 23373
Record Dates: First submitted 2009-05-21; First posted 2009-05-22 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2010-07

CONDITIONS: Vitiligo Vulgaris
Keywords: vitiligo; leucoderma
MeSH Terms: conditions — Vitiligo | interventions — Ginkgo Extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gingko biloba (Experimental): 60 mg of Ginkgo biloba (standardized to 15 mg ginkgofavonglycosides) given 2 times per day, with food, for 12 weeks.
  Interventions: Dietary Supplement: Ginkgo biloba

INTERVENTIONS:
Dietary Supplement: Ginkgo biloba — 60 mg Ginkgo biloba per capsule, standardized to 15 mg ginkgofavonglycosides per pill

SUMMARY:
Vitiligo is a common hypopigmentation disorder with significant psychological impact if occurring before adulthood. One study investigating the use of Ginkgo biloba for the treatment of vitiligo in adults reports effectiveness, but has significant flaws. We endeavor to conduct an open label pilot clinical trial replicating the previous trial on 12 adolescents 12 to 18 years old. The purpose of the pilot is to test the feasibility of recruitment and patient retention, variability of outcome measures, and identify major safety concerns. The pilot will use 60 mg of standardized G. biloba two times per day (BID) for 12 weeks. The primary outcome will be the validated Vitiligo European Task Force (VETF) evaluation form, secondary outcomes will include the Vitiligo Area Scoring Index (VASI), assess repigmentation via photographs, and will monitor and report adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* • males and females

  * 12 to 18 years old
  * self selected candidates identifying themselves to suffer with vitiligo vulgaris of any duration
  * minimum VASI score of 4, no maximum score (corresponding to a 3cm2 completely (100%) depigmented lesion, or a 6cm2 50% depigmented lesion)
  * stable or progressing vitiligo
  * mentally competent subjects able to adhere to the given protocol and treatments administered as interventions
  * normal on physical examination at the pre-study intake, and in the case of abnormalities the health care practitioner considers them to be clinically insignificant
  * written and informed consent
  * the potential candidate must have a family doctor that they have seen in the last 12 months
  * negative pregnancy test for menstruating women and if sexually active, a willingness to practice adequate birth control for the duration of the trial
  * diagnosis of vitiligo confirmed by supervising medical doctor

Exclusion Criteria:

* • use of medications contraindicated with Ginkgo biloba:

  * daily use of acetylsalicylic acid, ibuprofen, NSAIDs, fish oils, vitamin E
  * any prescription or use of blood thinners, anticoagulants, anti-platelet drugs, pentoxifylline, clotting factor replacements, antihypertensive medications, Thiazide diuretics, Acetylcholinesterase inhibitors, anticonvulsants, hypoglycemic agents, MAOI, SSRI, Nifedipine, Papaverine, Yohimgine, Sildenafil
  * history of diabetes, seizures, haemophilia
  * allergy or sensitivity to Ginkgo biloba or other constituents in the capsule
  * any treatment for vitiligo within the last 2 months
  * current use of Ginkgo biloba or within the last 2 months
  * mentally or physically incapacitated such that assent or informed consent cannot be obtained.
  * any history or other condition which the study physician regards as clinically significant to the study
  * a major illness considered to be clinically significant by the study physician within 2 months of the study start date
  * current participation in another intervention trial.
  * pregnancy or intent to become pregnant in the next 4 months
  * current alcoholism or substance abuse.
  * current history of tumors, any history of skin cancer
  * any current serious disorders determined to be clinically significant to the study.
  * breast feeding women
  * no prior skin grafts or surgeries, or scheduled surgeries of any kind.
  * any abnormalities on the INR, PTT, or CBC tests at baseline

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2009-05; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Vitiligo European Task Force assessment form | 12 weeks

SECONDARY OUTCOMES:
Vitiligo Area Scoring Index | 12 weeks
Health Canada - Canada Vigilence Adverse Reaction Form | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Orest Szczurko, ND MSc(cand), Principal Investigator — University of Toronto, Leslie Dan Faculty of Pharmacy; Heather Boon, PhD, Principal Investigator — University of Toronto, Leslie Dan Faculty of Pharmacy
Locations (1):
- Noumena Naturopathic Health Clinic, Mississauga, Ontario, Canada

REFERENCES:
- [Background] Parsad D, Pandhi R, Juneja A. Effectiveness of oral Ginkgo biloba in treating limited, slowly spreading vitiligo. Clin Exp Dermatol. 2003 May;28(3):285-7. doi: 10.1046/j.1365-2230.2003.01207.x. PMID 12780716
- [Derived] Szczurko O, Shear N, Taddio A, Boon H. Ginkgo biloba for the treatment of vitilgo vulgaris: an open label pilot clinical trial. BMC Complement Altern Med. 2011 Mar 15;11:21. doi: 10.1186/1472-6882-11-21. PMID 21406109
- See also: study recruitment website, providing study details, consent forms, etc — http://www.vitiligoresearch.org